CLINICAL TRIAL: NCT03876288
Title: Gastroparesis Outcome Longitudinal Database Enrolled Numerically
Acronym: GOLDEN
Status: Recruiting | Type: Observational
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Thomas Abell, The Arthur M Schoen MD Chair in Gastroenterology, University of Louisville
Other Study IDs: 13.0020
Record Dates: First submitted 2019-02-19; First posted 2019-03-15 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Immunotherapy; Immunoglobulins, Intravenous; Pyloromyotomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Laboratory testing, both clinical and research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- People presenting with the Sx of Gp: People presenting with the symptoms of gastroparesis. The three main interventions are GI neuromodulation, immunotherapy, and pyloric therapies.
  Interventions: Device: GI Neuromodulation; Drug: Immunotherapy; Procedure: Pyloric Therapies

INTERVENTIONS:
Device: GI Neuromodulation — The investigators would include follow up with: No treatment; temp GES only; temp followed by Perm GES; Other device therapies; specific pain therapies; drug therapies, including investigational drugs; immunotherapy; pyloric therapies; psychological/behavioral therapies; nutritional support; radiological and surgical therapies; infection rates related to procedures; if enrolled in any therapy research trials; morbidity and mortality after specific therapies; other treatments used.
  Other Names: Gastric electrical stimulation (GES)
Drug: Immunotherapy — The investigators would include follow up with: No treatment; temp gastric electrical stimulation (GES) only; temp followed by Perm GES; Other device therapies; specific pain therapies; drug therapies, including investigational drugs; immunotherapy; pyloric therapies; psychological/behavioral therapies; nutritional support; radiological and surgical therapies; infection rates related to procedures; if enrolled in any therapy research trials; morbidity and mortality after specific therapies; other treatments used.
  Other Names: Intravenous immunoglobulin
Procedure: Pyloric Therapies — The investigators would include follow up with: No treatment; temp gastric electrical stimulation (GES) only; temp followed by Perm GES; Other device therapies; specific pain therapies; drug therapies, including investigational drugs; immunotherapy; pyloric therapies; psychological/behavioral therapies; nutritional support; radiological and surgical therapies; infection rates related to procedures; if enrolled in any therapy research trials; morbidity and mortality after specific therapies; other treatments used.
  Other Names: Pyloromyotomy

SUMMARY:
GOLDEN is a longitudinal database of patients with the symptoms (Sx) of gastroparesis (Gp) who were seen and recorded at the University of Louisville from 2012 and is ongoing. Patients are enrolled and followed by sequential numbers and may include legacy patients seen at other centers by some of the same team and who are reported as part of the series. Outcome relate to patients Sx, survival, quality of life and other measures as detailed below, over time, regardless of whether any treatment was given or not. If treatments were administered GOLDEN allows for examination and stratification of outcome by groups both at baseline and at follow up.

DETAILED DESCRIPTION:
1. All patients seen with the Sx of Gp and who were evaluated for diagnosis and/or treatment
2. Including legacy patients who were seen and treated at previous locations (Mississippi, Arkansas, Tennessee) before Kentucky if they were part of a clinical research series.
3. Numbers of patients referred or consulted for Gp Sx who were Drug Refractory.
4. Interventions: GI Neuromodulation with gastric electrical stimulation (GES); Immunotherapy with Intravenous Immunoglobulin; Pyloric therapies such as pyloroplasty, surgical or endoscopic.
5. Data for evaluation by: Sx assessments by whatever scales used; Measures of health related quality of life; Psychological and pain assessments; Gastric emptying texts; Electrical measures including the following: single channel, low resolution and high resolution EGG, plus mucosal and serosal electrograms. High resolution EGG is also called Body Surface Mapping which is frequently measured in our patient population. ; Autonomic measure; Serologic measures; Full thickness biopsies; Measures of outpatient & Emergency Room Visits; Measures of hospitalization; Placement of endoscopic or surgical tubes; Radiological and Surgical procedures; Nutritional assessments; If enrolled in any research protocols for data; Stool biome measures; Metabolic measures; Other morbidity measures; Mortality

ELIGIBILITY:
Inclusion:

* Patients with the symptoms (Sx) of drug refractory gastroparesis
* Disordered nutrition by standardized assessment
* Ability to assess current symptom status
* Ability to measure other medical conditions

Exclusion:

* Anatomic obstruction of the GI Tract
* Pregnancy
* Inability of patient or guardian to sign informed consent, if needed
* Psychiatric disorders precluding assessment and treatment of the patient's GI condition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients seen
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Outcome GI Symptoms | Change from baseline to one week to one year
  The primary outcome measures are patient symptoms via the traditional gastroparesis patient reported outcome scale. It uses a 0-4 scale from none to worse on GI Symptoms; for example: Nausea,Vomiting, Anorexia/Early Satiety, Bloating/distension, Abdominal Pain. Scored as each item plus a total that is the sum of the individual scales.The five Sx subscales of 0-4 each are summed for a total score range 0-20

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Abell, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kasem F, Naing LY, Mathur P, McElmurray L, Moppins C, Daniels MW, Stocker A, Abell TL, Omer E. Patients With Gastroparesis Symptoms After Gastric Electrical Stimulation With and Without Tube Feedings. Neuromodulation. 2025 Nov 26:S1094-7159(25)00687-7. doi: 10.1016/j.neurom.2025.07.008. Online ahead of print. PMID 41307525
- [Derived] Kochar T, Cai W, Guardiola JJ, Mathur P, Hassan H, Atassi H, Stocker A, Hughes M, McElmurray L, Pinkston C, Abell TL. Nutritional Assessment in Patients after Gastric Electrical Stimulation (GES). J Clin Gastroenterol. 2024 Feb 1;58(2):136-142. doi: 10.1097/MCG.0000000000001826. PMID 36626193
- [Derived] Shine A, Mathur P, Ahmed S, Ramos S, McElmurray L, Stocker A, Pinkston C, Abell TL. Low-Resolution Electrogastrogram at Baseline and Response to Temporary Gastric Electrical Stimulation-A Comparison of Cutaneous With Mucosal Recordings. Neuromodulation. 2022 Dec;25(8):1150-1159. doi: 10.1016/j.neurom.2021.12.008. Epub 2022 Feb 17. PMID 35183451